CLINICAL TRIAL: NCT01310231
Title: A Randomized Phase II, Double Blind Trial of Standard Chemotherapy With Metformin (vs Placebo) in Women With Metastatic Breast Cancer Receiving First to Fourth Line Chemotherapy
Brief Title: A Trial of Standard Chemotherapy With Metformin (vs Placebo) in Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ozmosis Research Inc. (Industry)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OZM-027
Record Dates: First submitted 2011-02-18; First posted 2011-03-08 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Metformin
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): Metformin plus standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo and standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — metformin 850 mg bid in addition to standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Number of cycles: Until progression or unacceptable toxicity develops.
  Arms: Metformin
Drug: Placebo — Placebo bid in addition to standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Number of cycles: until progression or unacceptable toxicity develops.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the addition of metformin to standard chemotherapy improves progression free survival in women with metastatic breast cancer.

DETAILED DESCRIPTION:
A double blind Phase II randomized study of metformin versus (vs) placebo in non-diabetic women on first to fourth line chemotherapy with anthracycline, taxane, platinum, capecitabine or vinorelbine based regimens for metastatic or unresectable locally advanced breast cancer (BC). Patients were randomized to receive metformin 850 mg tablets or placebo once daily for two days as ramp-up, followed by one tablet twice a day for the duration of the study. Randomization was stratified by line of chemotherapy (1st, 2nd, 3rd and 4th line) and hormone receptor status (ER and/or PgR positive versus both negative). All patients were required to have measureable or non-measureable, but evaluable metastases at study entry. Metformin or placebo was to be continued until disease progression, even if chemotherapy was changed or stopped prior to disease progression. Recruitment took place at five sites in Ontario, Canada: Mount Sinai Hospital, Princess Margaret Cancer Centre, St. Michael's Hospital, Toronto and London Regional Cancer Centre, London.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive breast cancer with metastatic spread outside of breast, ipsilateral axillary and supraclavicular nodal areas (Histological confirmation of metastases is not required) OR, Locally advanced breast cancer that is refractory to initial anticancer treatment.
* A decision has been made to administer single or multiple agent first or second line chemotherapy that includes one of the following agents: anthracycline, taxane, platinum, capecitabine.
* Age: 18 to 75 years at the time of registration
* Invasive breast cancer, any ER or PgR status
* ECOG performance status 0-2
* Life expectancy of at least 6 months
* Adequate hepatic and renal function (SGOT and ALT < 1.8 X upper limit of normal for the institution, alkaline phosphatase ≤ 2X upper limit of normal for the institution, bilirubin within normal limits for the institution (expect in patients with Gilbert's syndrome who will be eligible regardless of bilirubin) and creatinine ≤ 130 umol/L)
* Blood counts: Neutrophils must be at least 1,000/mm3 and Platelets ≥ 75,000/mm3.
* Ability to understand and to provide written informed consent for the study
* Absence of any psychological, familial, sociological, or other patient related factors that might preclude compliance with the study protocol
* Measurable or non measurable (but evaluable) tumour must be present - radiologic or clinical evaluation must have been performed within 4 weeks prior to registration.

Exclusion Criteria:

* More than one previous line(s) of chemotherapy for metastatic disease - if prior chemotherapy has been administered, the last date of treatment must have been given at least 3 weeks prior to registration [any adjuvant systemic treatment is acceptable]
* If prior hormone therapy (as adjuvant or metastatic therapy) has been administered, it must have been stopped at least 3 weeks prior to registration
* Radiotherapy to a target or non target lesion within 4 weeks of registration
* Known CNS metastases
* History of cardiac failure
* Known hypersensitivity or allergy to metformin
* History of or known diabetes or baseline fasting glucose ≥ 7.0 mmol/L
* History of lactic or other metabolic acidosis
* Use of metformin within 3 months of registration
* Current or planned pregnancy or lactation in women of child-bearing potential. Patients of childbearing potential must have a negative serum pregnancy test.
* Fertile patients must agree to use an effective method of contraception while on study treatment; which could include IUD, condoms or other barrier methods of birth control
* Habitual alcohol intake of more than three drinks daily
* Concurrent use of any biguanide medication (other than metformin as a study medication)
* Patients with ≥ grade 2 diarrhea at baseline, malabsorption syndrome or unable to swallow oral medication
* Previous or concurrent malignancies, except non-melanoma skin cancers, unless curatively treated and with no evidence of recurrence for ≥ 5 years.
* Use of any investigational agent within 28 days prior to registration.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08-22 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Goodwin, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (5):
- Canada (5):
  - London Regional Cancer Program, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario

REFERENCES:
- [Result] Pimentel I, Lohmann AE, Ennis M, Dowling RJO, Cescon D, Elser C, Potvin KR, Haq R, Hamm C, Chang MC, Stambolic V, Goodwin PJ. A phase II randomized clinical trial of the effect of metformin versus placebo on progression-free survival in women with metastatic breast cancer receiving standard chemotherapy. Breast. 2019 Dec;48:17-23. doi: 10.1016/j.breast.2019.08.003. Epub 2019 Aug 22. PMID 31472446
- See also: Study Results — https://pubmed.ncbi.nlm.nih.gov/31472446/

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin plus standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Metformin: metformin 850 mg bid in addition to standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Number of cycles: Until progression or unacceptable toxicity develops.
- Placebo: Placebo and standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Placebo: Placebo bid in addition to standard chemotherapy (containing anthracyclines, platinum, taxanes or capecitabine; first or second line).
  Number of cycles: until progression or unacceptable toxicity develops.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 22 | 18
Received Intervention | 22 | 17
Discontinued Intervention | 0 | 1
Analyzed for Survival | 22 | 18
Analyzed for Response, Toxicity, QOL | 22 | 17
Completed | 22 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Full Range); unit: years] | 55 [39 to 75] | 57 [41 to 73] | 55.9 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Based on National Institutes of Health (NIH) Office of Management and Budget (OMB) Standards
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 5 | 4 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 17 | 13 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
ECOG Performance Scale [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Scale. Developed by the Eastern Cooperative Oncology Group, 1982 - Robert L. Comis, MD, Group Chair.
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG 0-1 | 20 | 16 | 36
    ECOG 2 | 2 | 2 | 4
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.5 [18.8 to 42.4] | 26.6 [20.5 to 37.9] | 26.5 [18.8 to 42.4]
Receptor Status [Number; unit: participants]
  (Estrogen Receptor (ER)/Progesterone Receptor (PR) positive | 19 | 15 | 34
  ER/PR negative | 3 | 3 | 6
Human epidermal growth factor receptor 2 (HER2) status [Number; unit: participants]
  HER2 positive | 2 | 4 | 6
  HER2 negative | 20 | 14 | 34
Any adjuvant chemotherapy [Number; unit: participants]
  Yes | 13 | 12 | 25
  No | 9 | 6 | 15
1st diagnosis to randomization [Mean (Full Range); unit: years] | 6.5 [0.1 to 24.6] | 4 [0.1 to 14.8] | 5.4 [0.1 to 24.6]
1st metastasis to randomization [Mean (Full Range); unit: years] | 0.8 [0 to 4.8] | 1.1 [0 to 5] | 0.9 [0 to 5]
Line of treatment [Number; unit: participants]
  1st line treatment | 15 | 12 | 27
  2nd line treatment | 4 | 3 | 7
  3+ lines treatment | 3 | 3 | 6
Any visceral disease [Number; unit: participants]
  Yes | 21 | 13 | 34
  No | 1 | 5 | 6
Involvement beyond bone and lymph nodes [Number; unit: participants]
  Yes | 22 | 15 | 37
  No | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival.
Description: Scans will be repeated every 9 weeks. Local follow up for survival will continue until all patients have died or for a maximum total follow up of 3 years, which ever occurs first. The two study arms will be compared in an intent to treat fashion using Cox proportional hazard analysis, with the stratification variables included in the model. Treatment discontinuation for toxicity or other reasons will be considered an event.
Time Frame: From date of randomization to first documented progression or death, which ever occurs first, assessed up to 3 years.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 18
months | 5.4 (1.04) | 6.3 (1.68)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Power: Final study plan called for 40 progression events, giving 80% power to detect a hazard ratio (HR) of 0.58 for PFS with a one-sided type I error of 20%, where the relatively high type I error reflects the Phase II status of the trial; Test type: Superiority; p = 0.71, Regression, Cox — One-sided p-value for group-effect obtained from Cox model. The prespecified threshold was 0.20 (one-sided); Cox model for PFS with metf/plac and the two randomization stratification variables line of chemotherapy and hormone receptor status; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.63 to 2.31] — Ratio of hazard of progression in the Metformin group relative to hazard in the Placebo group

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate in patients with measureable disease based upon RECIST Version 1.1. Patients will have scans repeated every 9 weeks and overall review of response across the study will be done every 6 months. The overall response rate is defined as number of patients with a best overall response of CR or PR, as a proportion of all patient with measurable disease at baseline. The response rate between arms will be compared using logistic regression with treatment as factor, adjusted for strata.
Time Frame: From baseline until time of best response, assessed up to 3 years
Population: Population is everyone with measurable disease (metformin 22, placebo 16)
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 16
Participants
  Clinical benefit | 12 | 7
  Progressive disease | 10 | 9
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.41, Regression, Logistic — Two-side p-value from a logistic regression model; Logistic regression model included metf/plac and the two stratification variables line of chemotherapy and hormone receptor status; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.45 to 6.99]

3. Secondary Outcome: Number of Participants With Grade 1 or 2 Adverse Events
Description: Adverse events graded using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
  Lower grade (grade 1 and 2) and higher grade (grade 3 and 4) are presented separately.
  A detailed breakdown of adverse events are given in the Adverse Events section
Time Frame: Up to 30 days after end of study
Population: Population is everyone who received study drug (metformin n=22, placebo n=17).
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 17
Participants | 15 | 6

4. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events
Description: as for outcome 3
Time Frame: Up to 30 days after end of study
Population: Population is everyone who received study drug (metformin n=22, placebo n=17).
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 22 | 17
Participants | 7 | 10

5. Secondary Outcome: EORTC Quality of Life Measures
Description: European Organization for Research and Treatment of Cancer (EORTC) quality of life measures: global health status and 5 functioning scales. Baseline and Cycle 2 outcomes are scaled from 0 to 100; higher scores indicate better functioning or better health status. CHANGE in these scales from baseline to cycle 2 is reported for each arm.
Time Frame: From baseline to cycle 2 of chemotherapy
Population: Population is everyone who completed BOTH baseline and Cycle 2 questionnaires (19 metformin, 16 placebo).
  3 metformin and 2 placebo patients did not complete the Cycle 2 EORTC questionnaire.
Measure: Mean (Standard Deviation); unit: EORTC functioning scale
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 19 | 16
EORTC functioning scale
  Global health Status | -12.7 (18.7) | 6.3 (19.6)
  Physical functioning | -6.0 (12.9) | 2.1 (12.1)
  Role functioning | -18.4 (27.7) | -2.1 (20.1)
  Emotional functioning | -2.6 (21.1) | 2.3 (16.7)
  Cognitive functioning | -0.9 (10.4) | 0 (17.2)
  Social functioning | -12.3 (29.8) | 4.2 (23.2)

6. Secondary Outcome: Change in Fasting Glucose (mmol/L)
Description: Change in fasting glucose from baseline to Cycle 2
Time Frame: Baseline to Cycle 2
Population: Population is everyone who had institutional glucose performed at BOTH baseline and Cycle 2 (19 metformin, 15 placebo).
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 7
mmol/L | -0.2 [-0.4 to 0.3] | 0 [-0.15 to 0.25]

7. Secondary Outcome: Change in Fasting Insulin
Description: Change in fasting insulin from baseline to Cycle 2
Time Frame: Baseline to Cycle 2
Population: Population is everyone who had sufficient fasting blood available for analysis at BOTH baseline and Cycle 2 (12 metformin, 7 placebo).
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 7
pmol/L | -7 [-14.25 to 0.5] | 1 [-13.5 to 20.5]

8. Secondary Outcome: Change in Insulin Resistance From Baseline to Cycle 2 Measured Using Homeostatic Model Assessment (HOMA-IR)
Description: HOMA-IR is an index calculated from fasting insulin (pmol/L) and glucose (mmol/L) as insulin/6.9 times glucose/22.5.
Time Frame: Baseline to Cycle 2
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 7
HOMA-IR score | -0.16 [-0.85 to 0] | 0.12 [-0.52 to 0.62]

9. Secondary Outcome: Immunohistochemical Predictors of Metformin Benefit and to Explore Changes in These Variables in Women Who Undergo Serial Biopsies of Their Metastases.
Description: Immunohistochemical analysis of different markers (IR, LKB1, phosphorylated AKT, S6K, ribosomal protein S6, 4E-BP1, and stathmin) pre and post first cycle of chemotherapy with metformin as well as in the original tumour tissue. Change in the phospho-markers of PI3K/mTOR will be summarized before and after the first cycle of chemotherapy with a focus on detection between the study arms.
Time Frame: Baseline and 3 weeks.
Population: Data not collected
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Gene Expression Predictors of Potential Metformin Benefit Including Exploration of Changes in These Variables in Women Who Undergo Serial Biopsies of Their Metastases
Description: Gene expression profiles in the baseline (original tumour) and, when available, pre and post cycle 1 chemotherapy will be established and change in gene signature pre and post chemotherapy will be explored.
Time Frame: Baseline and 4 weeks
Population: Data not collected
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The Adverse Events reporting period is defined as the time of consent signature until 30 days after date of off study treatment.
Description: All-cause mortality is available on all subjects (metformin n=22, placebo n=18). All the other Adverse Events are available on patients that received study drug (metformin n=22, placebo n=17).
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 19/22 | 15/18
Serious Adverse Events (participants affected / at risk) | 3/22 | 4/17
Other Adverse Events (participants affected / at risk) | 22/22 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=22) | Placebo (N=17)
febrile neutropenia with respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 1 (1) | 0 (0)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
febrile neutropenia with urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ascites with hyponatraemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
thromboembolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=22) | Placebo (N=17)
DIARRHOEA (Gastrointestinal disorders) | 16 | 7
NAUSEA (Gastrointestinal disorders) | 12 | 11
VOMITING (Gastrointestinal disorders) | 10 | 4
CONSTIPATION (Gastrointestinal disorders) | 5 | 8
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 | 6
DYSGEUSIA (Gastrointestinal disorders) | 5 | 4
FLATULENCE (Gastrointestinal disorders) | 3 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 3
DYSPEPSIA (Gastrointestinal disorders) | 4 | 1
STOMATITIS (Gastrointestinal disorders) | 2 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
FATIGUE (General disorders) | 11 | 7
HOT FLUSH (General disorders) | 3 | 2
PYREXIA (General disorders) | 2 | 3
MUCOSAL INFLAMMATION (General disorders) | 1 | 3
OEDEMA PERIPHERAL (General disorders) | 0 | 4
CHILLS (General disorders) | 1 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
LOCALISED OEDEMA (General disorders) | 0 | 2
PAIN (General disorders) | 0 | 2
ASTHENIA (General disorders) | 0 | 1
DYSGEUSIA (Nervous system disorders) | 5 | 4
PARAESTHESIA (Nervous system disorders) | 5 | 4
HEADACHE (Nervous system disorders) | 5 | 3
INSOMNIA (Nervous system disorders) | 2 | 3
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Nervous system disorders) | 4 | 1
VISION BLURRED (Nervous system disorders) | 3 | 2
DIZZINESS (Nervous system disorders) | 4 | 0
MUSCULAR WEAKNESS (Nervous system disorders) | 3 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1
HYPOAESTHESIA EYE (Nervous system disorders) | 0 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 7 | 6
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 4 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 1 | 1
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 1 | 3
RASH (Skin and subcutaneous tissue disorders) | 1 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 1
SKIN INFECTION (Skin and subcutaneous tissue disorders) | 1 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1
HOT FLUSH (Vascular disorders) | 3 | 2
DIZZINESS (Vascular disorders) | 4 | 0
EPISTAXIS (Vascular disorders) | 2 | 1
EMBOLISM (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
PHLEBITIS (Vascular disorders) | 0 | 1
PULMONARY EMBOLISM (Vascular disorders) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 6 | 2
OEDEMA PERIPHERAL (Metabolism and nutrition disorders) | 0 | 4
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
LOCALISED OEDEMA (Metabolism and nutrition disorders) | 0 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
DYSPNOEA (Cardiac disorders) | 1 | 6
DIZZINESS (Cardiac disorders) | 4 | 0
OEDEMA PERIPHERAL (Cardiac disorders) | 0 | 4
LOCALISED OEDEMA (Cardiac disorders) | 0 | 2
SKIN INFECTION (Infections and infestations) | 1 | 1
CYSTITIS (Infections and infestations) | 0 | 1
VISION BLURRED (Eye disorders) | 3 | 2
HYPOAESTHESIA EYE (Eye disorders) | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 2
NEUTROPHIL COUNT DECREASED (Investigations) | 3 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1
INSOMNIA (Psychiatric disorders) | 2 | 3
ANXIETY (Psychiatric disorders) | 1 | 2
DEPRESSION (Psychiatric disorders) | 0 | 1
MEMORY IMPAIRMENT (Psychiatric disorders) | 0 | 1
HOT FLUSH (Reproductive system and breast disorders) | 3 | 2
BREAST PAIN (Reproductive system and breast disorders) | 2 | 1
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 | 1
PHLEBITIS (Injury, poisoning and procedural complications) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
CYSTITIS (Renal and urinary disorders) | 0 | 1
POLLAKIURIA (Renal and urinary disorders) | 0 | 1
HYPERGLYCAEMIA (Endocrine disorders) | 2 | 0
HYPERSENSITIVITY (Immune system disorders) | 2 | 1
HEARING IMPAIRED (Ear and labyrinth disorders) | 0 | 1
SYNOVIAL CYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations include relatively small sample size, with associated imbalances in frequency of visceral (vs nonvisceral) metastatic disease, in HER2 positive and negative cancers, and in type of chemotherapy received in the metformin vs placebo arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No